CLINICAL TRIAL: NCT01917435
Title: Nasotracheal Intubation Assisted by a Video-stylet in Limited Mouth Opening Patient
Brief Title: Video-stylet for Nasotracheal Intubation in Limited Mouth Opening Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUH-IRB-20120254
Record Dates: First submitted 2013-07-10; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Anesthesia Intubation Complication
Keywords: fiberoptic bronchoscopy,; Video-stylet,; Nasotracheal Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fiberoptic bronchoscope (Experimental): Experimental: fiberoptic bronchoscope fiberoptic bronchoscope is used to facilitate for nasotracheal intubation.
  Interventions: Device: fiberoptic bronchoscope
- video-stylet (Experimental): Experimental: video-stylet video-stylet is used to facilitate for nasotracheal intubation.
  Interventions: Device: video-stylet

INTERVENTIONS:
Device: video-stylet
  Other Names: Device: video-stylet; Other Names:; The Clarus Video System
  Arms: video-stylet
Device: fiberoptic bronchoscope
  Other Names: fiberscope
  Arms: fiberoptic bronchoscope

SUMMARY:
The aim of the study is to investigate the efficiency of the Video-stylet (Trachway ®) and the fiberoptic bronchoscopy in facilitation of nasotracheal intubation in limited mouth opening patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-III
2. aged 20-65 years
3. Requiring Nasotracheal Intubation under general anesthesia
4. limited mouth open ,mouth open < 3 cm
5. unlimited neck motion

Exclusion Criteria:

1. Ankylosing arthritis patients.
2. BMI≧35 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
number of the patients with successful nasotracheal intubation and scoring modified intubation difficulty scale | half an hour
  Nasotracheal intubation is assisted by a video-stylet may be performed in patients undergoing Limited Mouth Opening following induction of anesthesia (fentanyl 2 micro-gram/kg, thiamylal 5 mg/kg) and is facilitated by cis-atracurium 0.2 mg/kg administration. propofol 1 mg/kg intravenously to blunt hemodynamic responses while intubation.
  a modified intubation difficulty scale to evaluate the difficulty of fiber-scope guided or trachway assisted nasotracheal intubation

SECONDARY OUTCOMES:
time to intubate | half an hour
  time of Intubating the nasotracheal tube (NT) from selected nostril to trachea is continuously calculated but separately into two parts. part one: from leaving off mask ventilation (mask removal from face), to the NT tip on the nasopharynx. part two: advancing NT from nasopharynx, through vocal cord into trachea, to present of 3 end tidal carbon dioxide waveforms.

OTHER OUTCOMES:
perioperative epistaxis, sore throat and hoarseness | 2 days
  Events of intubating related nasal bleeding are recorded on selected nostril and oral cavity at 3 minutes post-intubation and post-operatively. Incidences of sore throat and hoarseness are evaluated before patients out of recovery room and the following morning

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan